CLINICAL TRIAL: NCT04631276
Title: Clinical Study on Histamine H3 Receptor Occupancy of TS-091 by PET Examination in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS091-1402
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single evaluation of H3 receptor occupancy (Experimental): Subjects received single-dose of 0.1, 0.2, 0.4, 1, 2.5, 25 mg TS-091 prior to an evaluation of H3 recepto occupancy
  Interventions: Drug: TS-091
- Multiple evaluations of H3 receptor occupancy (Experimental): Subjects received single-dose of 5, 12.5, 25 mg TS-091 prior to Multiple evaluations of H3 recepto occupancy
  Interventions: Drug: TS-091

INTERVENTIONS:
Drug: TS-091 — Subjects received single-dose of 0.1, 0.2, 0.4, 1, 5, 12.5 and 25 mg of TS-091 (tablets or drug substance powder)

SUMMARY:
To evaluate the following items by PET examination in Japanese heathy adult male subjects who received single oral administration of TS-091 in an unblinded manner.

1. Relationship between plasma concentration and H3 receptor-occupancy of TS-091
2. Time course changes in H3 receptor-occupancy of TS-091

ELIGIBILITY:
Inclusion Criteria:

Subjects who met all of the following criteria.

* Age: between ≥20 years and <40 years at the time of providing written consent for participation in the study.
* Body mass index (BMI): ≥18.5 and <25.0 on the day of screening test.
* Subject who received a prior explanation on the study and was able to understand its content and capable of providing voluntary written consent for participation in the study.
* Other protocol defined inclusion criteria could apply-

Exclusion Criteria:

Subjects who came under any of the following exclusion criteria.

* Subjects who were considered to have some disease and not healthy by the investigator or subinvestigator according to his medical judgment based on the results of screening test
* Subjects with a drug or food allergy or a history thereof.
* Subjects with a significant allergic disposition (e.g. asthma requiring treatment) or a history thereof.
* Subjects with a history of heparin-induced thrombocytopenia.
* Other protocol defined exclusion criteria could apply

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2015-12-16 (Actual); Study Completion 2015-12-16 (Actual)

PRIMARY OUTCOMES:
H3 receptor occupancy | 2 hours after administration of TS-091
  H3 receptor occupancy is calcurated at 2 hours after administration of TS-091.
Changes in the H3 receptor occupancy | 2, 6, and 26 hours after administration of TS-091
  Changes in the H3 receptor occupancy is calcurated at 2, 6, and 26 hours after administration of TS-091
Plasma concentration of unchanged TS-091 | 2, 6, and 26 hours after administration of TS-091
  Plasma concentration of unchanged TS-091 is calcurated at 2, 6, and 26 hours after administration of TS-091

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kimura Y, Takahata K, Shimazaki T, Kitamura S, Seki C, Ikoma Y, Ichise M, Kawamura K, Yamada M, Zhang MR, Higuchi M, Nishino I, Suhara T. Pharmacokinetic and pharmacodynamic assessment of histamine H3 receptor occupancy by enerisant: a human PET study with a novel H3 binding ligand, [11C]TASP457. Eur J Nucl Med Mol Imaging. 2022 Mar;49(4):1127-1135. doi: 10.1007/s00259-021-05571-1. Epub 2021 Oct 15. PMID 34651222